CLINICAL TRIAL: NCT03920930
Title: Optimization of a Fast-track Concept for Knee Replacement: A Single-blind, Randomized, Controlled Clinical Trial
Brief Title: Optimization of a Fast-track Concept for Knee Joint Replacement
Acronym: KneeOptOut2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Sascha Treskatsch, Prof. Dr. med., Head of Department, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KneeOptOut2
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Knee Arthropathy; Postoperative Pain; Postoperative Complications
Keywords: ERAS; pain; knee arthroplasty; joint pain; regional anaesthesia
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications; Pain; Arthralgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Investigator and treating physicians are different in this trial, that means, the assessor of primary study endpoint will be blinded regarding group allocation. Patients receive either early or late local infiltration technique perioperatively. Patients will be blinded against early or late local infiltration technique. Blinding of the treating physician will not be possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early-intraoperative Local infiltration technique (Experimental): A distal regional anaesthesia is performed in which the nerves are blocked by a local anaesthetic in the tissue in the immediate vicinity of the operating area ("tissue infiltration technique"). The LIA is applied in a total of 4 steps during the preparation of the knee joint: 1. after the skin incision, 2. after the capsule incision, 3. after complete exposure of the knee joint, 4. when the posterior knee capsule is reached.
  Interventions: Procedure: Early local infiltration analgesia
- Late-intraoperative Local infiltration technique (Active Comparator): A distal regional anaesthesia is performed in which the nerves are blocked by a local anaesthetic in the tissue in the immediate vicinity of the operating area ("tissue infiltration technique"). The LIA is applied after the preparation of the femur and tibia bone shortly before the prosthesis is inserted and during the retreat from the knee joint.
  Interventions: Procedure: Late local infiltration analgesia

INTERVENTIONS:
Procedure: Late local infiltration analgesia — Patient receive an infiltration of local anaesthetics around the knee directly after total knee replacement for postoperative pain control.
  Other Names: late LIA
  Arms: Late-intraoperative Local infiltration technique
Procedure: Early local infiltration analgesia — The local infiltration analgesia is applied in a total of 4 steps during the preparation of the knee joint: 1. after the skin incision, 2. after the capsule incision, 3. after complete exposure of the knee joint, 4. when the posterior knee capsule is reached.
  Other Names: early LIA
  Arms: Early-intraoperative Local infiltration technique

SUMMARY:
In an estimated 150,000 patients, a knee joint replacement is performed in Germany every year. The perioperative care of the patients aims at an optimal surgical technique, which leads to a high functionality in the joint, and above all at an adequate pain treatment. Patients experience pain especially intraoperatively and in the first days after the operation. The intensity of pain is a decisive factor that can hinder the patient's mobilization. In the KneeOptOut study (ethics application number EA4/009/17), which has already been successfully carried out and approved by this ethics committee, it was shown that the use of local infiltration anaesthesia (LIA) for pain therapy after primary knee endoprosthetics is comparable to catheter-supported regional anaesthesia (manuscript under review at the European Journal of Anaesthesiology). During surgery, the morphine requirement of patients in the LIA group was significantly higher than that of patients who underwent catheterization. Postoperatively, however, both subjective pain by VAS and opiate consumption were comparable.

In order to optimize the intraoperative opiate need/consumption, an early-intraoperative procedure for local infiltration anesthesia will now be compared with the previous late-intraoperative procedure. Both procedures correspond to SOP for the treatment of primary knee endoprostheses and are currently used depending on the surgeon's requirements.

ELIGIBILITY:
Inclusion Criteria:

• patients undergoing elective, primary knee joint replacement in combined general anaesthesia

Exclusion Criteria:

* heart insufficiency NYHA >2
* liver insufficiency > CHILD B
* evidence of diabetic polyneuropathy
* severe adipositas BMI >40
* patients < 18 years
* pregnancy
* in case of police custody
* participation in a paralleled interventional RCT in a time frame of 30 days
* chronic opioid therapy >3 months before scheduled surgery
* allergy against medication required for surgery or anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | intraoperative, up to 3 hours
  amount of opioids administered intraoperative measured as equivalent dose to morphin

SECONDARY OUTCOMES:
time to first mobilisation (standing) | up to 48 hours postoperatively
  time from end of surgery until patients is able to stand
patients satisfaction (11-point likert scale) | up to 7 days postoperatively
  global satisfaction of patients
time to first mobilisation (walking) | up to 7 days postoperatively
  time from end of surgery until patients is able to walk
time to achieve full joint mobility | up to 7 days postoperatively
  time to achieve full joint mobility (0/0/90°)
Janda grade of both legs at first day after surgery | up to 24h postoperatively
  best Janda grade in both legs the day after surgery
Pain intensity | up to 7 days postoperatively
  intensity of pain in all patients meausered by numeric rating scale (NRS)
rescue pain medication | up to 7 days postoperatively
  number of patients requiring rescue pain medication
time to discharge | up to 14 days postoperatively
  time to discharge from hospital
Opioid consumption (hospital) | up to 14 days postoperatively
  amount of opioids administered until discharge measured as equivalent dose to morphin
delirium | up to 7 days postoperatively
  incidence of postoperative delirium measured by Nursing Delirium Screening Scale (NuDeSc)
postoperative nausea and vomiting (PONV) | up to 7 days postoperatively
  incidence of PONV
surgeon satisfaction (6-point likert scale) | intraoperative, up to 3 hours
  satisfaction of surgeon in points of clarity of the operative field, change of the operative field by LIA and overall satisfaction represented in one value

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Background] Morin AM, Wulf H. [High volume local infiltration analgesia (LIA) for total hip and knee arthroplasty: a brief review of the current status]. Anasthesiol Intensivmed Notfallmed Schmerzther. 2011 Feb;46(2):84-6. doi: 10.1055/s-0031-1272875. Epub 2011 Feb 10. German. PMID 21312140
- [Background] Perret M, Fletcher P, Firth L, Yates P. Comparison of patient outcomes in periarticular and intraarticular local anaesthetic infiltration techniques in total knee arthroplasty. J Orthop Surg Res. 2015 Jul 31;10:119. doi: 10.1186/s13018-015-0249-x. PMID 26227482
- [Background] Peters CL, Shirley B, Erickson J. The effect of a new multimodal perioperative anesthetic regimen on postoperative pain, side effects, rehabilitation, and length of hospital stay after total joint arthroplasty. J Arthroplasty. 2006 Sep;21(6 Suppl 2):132-8. doi: 10.1016/j.arth.2006.04.017. PMID 16950075
- [Background] Suthersan M, Pit S, Gordon L, Loman M, Pezzutti B, Freihaut R. Local infiltration analgesia versus standard analgesia in total knee arthroplasty. J Orthop Surg (Hong Kong). 2015 Aug;23(2):198-201. doi: 10.1177/230949901502300217. PMID 26321550
- [Background] Kastelik J, Fuchs M, Kramer M, Trauzeddel RF, Ertmer M, von Roth P, Perka C, Kirschbaum SM, Tafelski S, Treskatsch S. Local infiltration anaesthesia versus sciatic nerve and adductor canal block for fast-track knee arthroplasty: A randomised controlled clinical trial. Eur J Anaesthesiol. 2019 Apr;36(4):255-263. doi: 10.1097/EJA.0000000000000929. PMID 30562225